CLINICAL TRIAL: NCT04674748
Title: A Phase 1 Study Exploring the Safety, Tolerability, and Pharmacokinetics of INCB086550 in Japanese Participants With Advanced Solid Tumors
Brief Title: To Assess the Safety, Tolerability and Pharmacokinetics of INCB086550
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated early due to a business decision.
Sponsor: Incyte Biosciences Japan GK (Industry)
Responsible Party: Sponsor
Organization: Incyte Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 86550-104
Record Dates: First submitted 2020-12-07; First posted 2020-12-19 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumors
Keywords: Advanced; Metastatic; Refractory; Relapsed
MeSH Terms: conditions — Neoplasm Metastasis; Recurrence

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dose Escalation of INCB086550 (Experimental): In this study 3 dose levels will be evaluated to determine the MTD or RP2D (Decided by SMC according to the safety and PK data)
  Interventions: Drug: INCB086550

INTERVENTIONS:
Drug: INCB086550 — Each Participant will be treated at the specified dose level with a minimum of 3 subjects at each dose level. After the RP2D of INCB086550 is identified, the dose level will be expanded to better characterize the safety and tolerability and PK.

SUMMARY:
This study will assess the safety, tolerability, and PK of INCB086550 and determine the Maximum Tolerated Dose (MTD) and/or recommended Phase 2 Dose(RP2D) of INCB086550, whichever is lower, in Japanese participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to conform to and comply with all Protocol requirements, including all scheduled visits, Protocol procedures, and the ability to swallow oral medication.

  * Histologically or cytologically confirmed diagnosis of any locally advanced or metastatic solid tumors with measurable lesions per RECIST v1.1 not amenable to local or other curative therapy.
  * Disease progression after treatment with available therapies that are known to confer clinical benefit or intolerant to or ineligible for standard treatment.
  * ECOG performance status of 0 or 1.
  * Life expectancy > 12 weeks.
  * Female participants should agree to use medically acceptable contraceptive measures should not be breastfeeding, and must have a negative pregnancy test before the start of study drug administration if of childbearing potential.
  * Female participants of childbearing potential must understand and accept that pregnancy must be avoided during participation in the study, from screening through 90 days after the last dose of study drug.

Male participants should avoid unprotected sex with women of childbearing potential during the study and for a washout period of 90 days after the last dose of study drug.

* For participants who will be enrolled in the study and receive the RP2D of INCB086550 in the expanded cohort: Willingness to undergo a tumor biopsy to obtain tumor tissue. Pretreatment and on-treatment tumor biopsies are required.

Exclusion Criteria:

* Laboratory values not within the Protocol-defined range.
* Clinically significant cardiac disease, including left ventricular ejection fraction < 40%, unstable angina, acute myocardial infarction within 6 months of Cycle 1 Day 1, New York Heart Association Class III or IV congestive heart failure, and arrhythmia requiring therapy.
* History or presence of abnormal ECG that, in the investigator's opinion, is clinically meaningful.
* Untreated brain or CNS metastases or brain or CNS metastases that have progressed (eg, evidence of new or enlarging brain metastasis or new neurologic symptoms attributable to brain or CNS metastases).
* Active or inactive autoimmune disease or syndrome (eg, rheumatoid arthritis, moderate or severe psoriasis, multiple sclerosis, inflammatory bowel disease) that has required systemic treatment in the past 2 years or receiving systemic therapy for an autoimmune or inflammatory disease (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs).
* Diagnosis of immunodeficiency or receiving chronic systemic steroid therapy (doses exceeding 10 mg daily of prednisolone equivalent) or any other form of immunosuppressive therapy within 7 days before the first dose of study drug. Use of short courses of steroids for procedure prophylaxis, inhaled or topical steroids, or systemic corticosteroids ≤ 10 mg is permitted.
* Known additional malignancy that is progressing or requires active treatment.
* Evidence or a history of interstitial lung disease or active, noninfectious pneumonitis.
* Treatment with anticancer medications or investigational drugs is prohibited within the following intervals before the first administration of study drug.
* Concomitant treatment with moderate and potent CYP3A4/CYP3A5 inhibitors or inducers.
* Receipt of a live vaccine within 3 months of the first dose of study drug.
* Active infection requiring systemic therapy.
* Systemic antibiotic therapy. A washout of 28 days is required before the first dose of INCB086550.
* Probiotic supplement usage during screening and throughout the study treatment period.
* Known active HBV or HCV infection or risk of reactivation of HBV or HCV.
* History of organ transplant, including allogeneic stem cell transplantation.
* Known hypersensitivity or severe reaction to any component of study drug or formulation components.
* Inability to swallow food or any condition of the upper gastrointestinal tract that precludes administration of oral medications.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* Inability or unlikeliness of the participant to comply with the dose schedule and study evaluations, in the opinion of the investigator.
* Inadequate recovery from toxicity and/or complications from a major surgery before starting therapy.
* Women who are pregnant or breastfeeding.
* Inability of the participant (or parent, guardian, or legally authorized representative) to comprehend the ICF or unwillingness to sign the ICF.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAE) | Up to 27 months
  Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug/treatment.

SECONDARY OUTCOMES:
Objective Response Rate | Up to 2 years
  Defined as the percentage of participants with best overall response of CR or PR as determined by the investigator per RECIST v1.1.
Cmax | Pre dose,Post dose on Cycle 1 Day 1 & Day 15, Pre dose on Cycle 1 Day 8, Cylce 2 Day 21, and Cycle 3 Day 1 (each cycle 28 days)
  Maximum Observed Plasma concentration of INCB086550
Tmax | Pre dose,Post dose on Cycle 1 Day 1 & Day 15, Pre dose on Cycle 1 Day 8, Cylce 2 Day 21, and Cycle 3 Day 1 (each cycle 28 days)
  Time to reach maximum (peak) Plasma concentration of INCB086550
Cmin | Pre dose,Post dose on Cycle 1 Day 1 & Day 15, Pre dose on Cycle 1 Day 8, Cylce 2 Day 21, and Cycle 3 Day 1 (each cycle 28 days)
  Trough plasma concentration of INCB086550
AUC0-t | Pre dose,Post dose on Cycle 1 Day 1 & Day 15, Pre dose on Cycle 1 Day 8, Cylce 2 Day 21, and Cycle 3 Day 1 (each cycle 28 days)
  Area under the single-dose plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration of INCB086550
AUC0-∞ | Pre dose,Post dose on Cycle 1 Day 1 & Day 15, Pre dose on Cycle 1 Day 8, Cylce 2 Day 21, and Cycle 3 Day 1 (each cycle 28 days)
  area under the single-dose plasma concentration-time curve from Hour 0 to infinity of INCB086550
AUC(0-τ) | Pre dose,Post dose on Cycle 1 Day 1 & Day 15, Pre dose on Cycle 1 Day 8, Cylce 2 Day 21, and Cycle 3 Day 1 (each cycle 28 days)
  AUC to the end of dosing period of INCB086550
t1/2 | Pre dose,Post dose on Cycle 1 Day 1 & Day 15, Pre dose on Cycle 1 Day 8, Cylce 2 Day 21, and Cycle 3 Day 1 (each cycle 28 days)
  Terminal half-life of INCB086550
CL/F | Pre dose,Post dose on Cycle 1 Day 1 & Day 15, Pre dose on Cycle 1 Day 8, Cylce 2 Day 21, and Cycle 3 Day 1 (each cycle 28 days)
  Oral dose clearance of INCB086550
λz | Pre dose,Post dose on Cycle 1 Day 1 & Day 15, Pre dose on Cycle 1 Day 8, Cylce 2 Day 21, and Cycle 3 Day 1 (each cycle 28 days)
  Terminal elimination rate constant of INCB086550
Vz/F | Pre dose,Post dose on Cycle 1 Day 1 & Day 15, Pre dose on Cycle 1 Day 8, Cylce 2 Day 21, and Cycle 3 Day 1 (each cycle 28 days)
  Apparent oral dose volume of distribution of INCB086550

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - National Cancer Center Hospital - East, Chiba
  - National Cancer Center Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency